CLINICAL TRIAL: NCT06488443
Title: Randomized Control Study to Study the Effect of Yoga on Reducing Craving in Tobacco Dependent Individuals Who Want to Quit Tobacco Use
Brief Title: Effect of Yoga on Reducing Craving in Tobacco Dependent Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); St.John's Medical College and Hospital (Unknown)
Responsible Party: Principal Investigator, Vishwajit Nimgaonkar, MD PhD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY23050176; D43TW009114 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-07-05 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Tobacco Dependence
Keywords: Tobacco dependence; Smoking; Craving; Fagerstorm test
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: The proposed study is a Randomized controlled trial.. It is two arm study, intervention arm and control arm. Intervention arm will be imparted yoga while control arm will be given the WHO 5As model intervention.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to the randomisation. Principal investigator will not be involved in randomization of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-yoga (Experimental): Participants in intervention arm will receive intervention from an instructor who would be trained in the intervention by the yoga adviser. One week of yoga intervention with the first session offline and the rest of the 6 sessions online
  Interventions: Behavioral: Yoga
- WHO 5As model intervention (Active Comparator): The control group will be given the WHO 5As model intervention to help patients ready to quit.
  Interventions: Behavioral: WHO 5As model intervention

INTERVENTIONS:
Behavioral: Yoga — Participants in yoga arm will receive intervention from an instructor who would be trained in the intervention by the yoga adviser.All the yoga exercises selected for this study are low-impact and involve highly controlled movements. All yoga exercises will be taught and supervised by a skilled yoga-instructor. The yoga-instructor will take great care to emphasize to participants that they should not go beyond their usual range of motion/comfort for any of the yoga exercises.
  Arms: Intervention-yoga
Behavioral: WHO 5As model intervention — WHO 5As model to help patients ready to quit. The five major steps to intervention are the "5 A's": Ask, Advise, Assess, Assist, and Arrange.
  Arms: WHO 5As model intervention

SUMMARY:
Yoga is a culturally acceptable practice that can reduce craving and help people quit tobacco. There is a need to evaluate the feasibility of implementation of a well- designed yoga protocol to address craving in individuals who use tobacco in India.

DETAILED DESCRIPTION:
There is a high prevalence of tobacco use in the community that continue to remain underserved in terms of intervention and support for their tobacco use. Yoga is a culturally acceptable practice that can reduce craving and help people quit tobacco. However, we didn't come across Indian studies looking at yoga to reduce craving in individuals who use tobacco. There is a need to evaluate the feasibility of implementation of a well- designed yoga protocol to address craving in individuals who use tobacco in India.

Aim: To study the feasibility of yoga in reducing craving in individuals who use tobacco

Objectives:

Primary

* To evaluate the feasibility of yoga based intervention on craving in tobacco dependent individuals who want to quit tobacco use Secondary/tertiary
* To assess the effect on abstinence
* To assess quit rate

Sampling frame:

Screened positive participants will be recruited from Rural community health and training centre, Mugalur, Tobacco cessation centre and OPDs of Department of general medicine, pulmonary medicine, cardiology, oncology, ENT and dental surgery and other super speciality OPD at SJMCH

.

Sample recruitment/sampling method:

Participants who fulfilled the inclusion criteria will be approached by the principal investigator and/or junior research fellow, and those who agreed to participate in the study will be randomly allocated to one of two groups via simple randomization. Randomisation will be computerised. This will be done in blocks of 10. Outcome assessor will be blinded to the randomisation. Principal investigator will not be involved in randomization of participants.

Training/ interventions/assessments/ procedures in the study -Participants in yoga arm will receive intervention from an instructor who would be trained in the intervention by the yoga adviser.

Procedure:

Screening positive participants fulfilling eligibility criteria, information regarding study is given and informed consent is documented. Selection of a quit date within 21 weeks.

Standard of living index(SLI) or Modified Kuppuswamy Scale for sociodemographic data (10mins), Fagerstrom scale(5 mins), Motivation to stop smoking (1 min) .

Participants are randomized into intervention and TAU groups with 48 participants each.

For intervention group, sixty minute yoga session will be imparted. The first session shall be offline, the rest of the 6 sessions shall be online.. After Completion all assessments will be done again both of intervention and TAU groups.Follow up at 21 weeks, 1 month and at 3 months.

-To assess relapse

Hypothesis Yoga will be a feasible method to reduce craving in tobacco dependent individuals who want to quit tobacco use

ELIGIBILITY:
Inclusion Criteria:

* -Tobacco dependent individuals (Fagerstrom test for tobacco dependence score more than or equal to 4)

  * -Men aged 18 to 65 years
  * -Recruited from Rural community health and training centre, Mugalur, Tobacco cessation centre and OPDs of Department of general medicine, pulmonary medicine, cardiology, oncology, ENT and dental surgery and other superspeciality OPD at SJMCH

Exclusion Criteria:

Patients with recent alcohol use (last 3 months) and use of other drugs of abuse

* -Patients with clinical diagnosis of Intellectual disability
* -Comorbid Major mental illness including Dementia, Psychosis, Recurrent depressive disorder, Bipolar affective disorder, OCD, generalized anxiety disorder, Panic disorder and Phobias, diagnosed within the last 6 months.
* -Patients with recent MI and stroke in the last 3 months or those physically unable to perform the yoga postures due to physical disabilities determined by clinical interview.

  * -Patients with severe hypertension(SBP≥180mmHg and BP≥120mmHg)
  * -Patients with seizures disorder
  * -Patients with COPD(GOLD-2,3 and 4)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of yoga based intervention | After one week of intervention
  To evaluate the feasibility of yoga-based intervention in changing craving of tobacco in comparison to WHO 5As intervention on individuals who want to quit tobacco use with Visual Analogue scale (upto score 3 not useful: scores 4,5,6 neutral; 7,8,9, 10 useful) Minimum score is 0 and maximum score is 10
Craving of tobacco after intervention | After one week of intervention
  To evaluate the feasibility of yoga-based intervention in changing craving of tobacco measured by Brief Questionnaire of Smoking Urges in comparison to WHO 5As intervention on individuals who want to quit tobacco use using (Scale is 10 items likert scale and total of all item scores is the score, more the score more is the craving)Minimm score is 0 and maximum is 100.
Craving of tobacco one month follow up | 1 month after intervention
  To evaluate the feasibility of yoga-based intervention in changing craving of tobacco measured by Brief Questionnaire of Smoking Urges in comparison to WHO 5As intervention on individuals who want to quit tobacco use (Scale is 10 items likert scale and total of all item scores is the score, more the score more is the craving) Minimum score is 0 and maximum is 100.
Craving of tobacco three months follow up | 3 months after intervention
  To evaluate the feasibility of yoga-based intervention in changing craving of tobacco (Scale is 10 items likert scale and total of all item scores is the score, more the score more is the craving)measured by Brief Questionnaire of Smoking Urges in comparison to WHO 5As intervention on individuals who want to quit tobacco use. The minimum score is 0 and maximum score is 100.

SECONDARY OUTCOMES:
Relapse rate of tobacco use (Number of participants start using tobacco again) | After one week of intervention
  To compare effect of yoga Relapse rate of tobacco use on abstinence with WHO 5As intervention group
Relapse rate of tobacco use(One month sustainability) ((Number of participants start using tobacco again) | 1 month after intervention
  To compare effect of yoga intervention on relapse rate of tobacco use with WHO 5As intervention group
Relapse rate of tobacco use (Three months sustainability)(Number of participants start using tobacco again) | 3 months after intervention
  To compare effect of yoga intervention on relapse rate of tobacco use with WHO 5As intervention group
Quit rate of tobacco | After one week of intervention
  To compare the change in quit rate after yoga intervention with WHO 5As intervention group
Quit rate of tobacco (One month sustainability) | 1 month after intervention
  To compare the change in quit rate after yoga intervention with WHO 5As intervention group
Quit rate of tobacco (Three month sustainability) | 3 months after intervention
  To compare the change in quit rate after yoga intervention with WHO 5As intervention group
Relapse rate of smoking | After one week of intervention
  To compare the change in relapse rate after yoga intervention with that of WHO 5As intervention group
Relapse rate of smoking (One month sustainability) | 1 month after intervention
  To compare the change in relapse rate after yoga intervention with that of WHO 5As intervention group
Relapse rate of smoking (Three month sustainability) | 3 months after intervention
  To compare the change in relapse rate after yoga intervention with that of WHO 5As intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit Nimgaonkar, MD, PhD, Principal Investigator — University of Pittburgh
Locations (1):
- St.John's Medical College and Hospital, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: One year after publication of this study.
Access Criteria: For individual participant data, meta-analysis.